CLINICAL TRIAL: NCT02022787
Title: Value of Various Chemokines in the Detection and Follow up of RCC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Boris Friedman, MD, Carmel Medical Center
Other Study IDs: CMC-13-0064-CTIL; CMC-13-0064 (Registry Identifier: Title: Chemokines and RCC)
Record Dates: First submitted 2013-10-30; First posted 2013-12-30 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Clear Cell Renal Cell Carcinoma
Keywords: RCC; Chemokines; nephrectomy; partial nephrectomy
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Renal tumor tissue and patients' serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Renal cell carcinoma: Patients with renal cell carcinoma scheduled for partial or radical nephrectomy
  Interventions: Other: patients with renal cell carcinoma

INTERVENTIONS:
Other: patients with renal cell carcinoma — Chemokines that may be elevated in patients with RCC

SUMMARY:
This study was designed as a pilot study to try and find a Chemokine that may be specific for renal cell carcinoma

DETAILED DESCRIPTION:
I n previous studies that were initiated in experimental models of different inflammatory autoimmune diseases and then extended to humans, we have shown that in the course of inflammatory autoimmune diseases, the immune system selectively generates an auto-Ab response to a few inflammatory mediators, mostly chemokines and cytokines, which are thought to participate in promoting the inflammatory process (1-6). For example, we showed that patients suffering from rheumatoid arthritis (RA) but not osteoarthritis display a significant level of neutralizing auto- Abs directed against TNF-a (tumor necrosis factor)(3). These patients did not mount any auto-Ab response either to several key inflammatory chemokines or to regulatory mediators, such as IL-10(interleukin-10) or TGF-b(tumor growth factor)(, or even the chemokine CXCL12(C-X-C motif chemokine 12), which also functions as a regulatory mediator that selects Ag-specific IL-10-producing CD4+(cluster of differentiation 4) T cells (7).

Complementary experiments suggested that in experimentally induced RA, these anti-TNF-a auto-Abs participate in the natural regulation of disease and restrain-although they are incapable of totally preventing-its development (3). Nevertheless, their selective amplification by targeted DNA vaccines led to rapid recovery from an ongoing disease (8). These studies also showed that selective breakdown of tolerance to TNF-a is due to its preferential expression at a partially immune-restricted site undergoing a destructive process (3, 8). Very recently, we have shown that type I diabetes mellitus (T1DM) patients preferentially display auto-Ab production to CCL3( Chemokine (C-C motif) ligand 3) and not to several other proinflammatory chemokines (9).

It is yet to be proven that this chemokine dominates the chemokine expression at the autoimmune site. Nevertheless, a previous study showing that selective neutralization of CCL3 suppresses T1DM in NOD mice has implications for the important role of this chemokine in this disease (10). Similarly to organ-specific autoimmunity in various cancer diseases, one of which is cancer of the prostate (CaP), key inflammatory chemokines are expressed at the primary tumor site, which also undergoes a destructive process at a restricted site. In a previous study we showed that in primary tumor sections of prostate cancer subjects, CCL2Chemokine (C-C motif) ligand 2) is predominantly expressed at the tumor site over other chemokines that also have been associated with tumor development, including: CXCL12, CXCL10, CXCL8, CCL3,CCL4, and CCL5. Subsequently, the immune response selectivity mounts an Ab-based response to CCL2. These Abs are neutralizing Abs. These findings hold diagnostic and therapeutic implications.

Little is known about the possible function of chemokine receptors in the development and progression of renal cell carcinoma (RCC). Few studies exist dealing with gene expression of chemokines in RCC. We therefore suggest a study checking antibody response to a few chemokines

ELIGIBILITY:
Inclusion Criteria:

Patients with renal cell carcinoma of one or both kidneys scheduled for surgical resection

-

Exclusion Criteria:

Males with elevated PSA (prostatic specific antigen ) Any other untreated malignancy -

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for partial or radical nephrectomy
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Measurement of the titers of chemokines before and after tumor resection | before nephrectomy (day of surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Avi Stein, M.D., Principal Investigator — Carmel Medical Center
Locations (1):
- Carmel Medical Center, Haifa, Israel